CLINICAL TRIAL: NCT01054209
Title: A Study to Determine the Effectiveness of a Warming Mattress in Preventing Inadvertent Peri-operative Hypothermia and Shivering in Patients Undergoing Elective Cesarean Section
Brief Title: Electric Warming Mattress to Prevent IPH During LSCS
Acronym: ObsIPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dr C. Mark Harper, Consultant Anaesthetist, Brighton and Sussex University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09/165/HAR
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Hypothermia; Anesthesia; Obstetric Anesthesia Problems
Keywords: Inadvertent Peri-operative Hypothermia; Shivering; Caesarean Section; Elective; Warming Mattress; Regional Anaesthesia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: standard care, no warming (No Intervention): Control arm. Full standard care. No mattress warming. May receive warmed fluids if standard practise for clinician
- B: electric warming mattress (Active Comparator): Warming with warming mattress
  Interventions: Device: Warming with warming mattress

INTERVENTIONS:
Device: Warming with warming mattress — Reusable pressure relieving warming mattress. Principle use is to warm patients to prevent hypothermia peri-operatively.
  Inditherm Alpha systems, OTM1: 1900mm x 585mm
  Other Names: Inditherm Alpha systems, OTM1: 1900mm x 585mm
  Arms: B: electric warming mattress

SUMMARY:
This study will demonstrate whether an electric warming mattress can reduce the number of patients who get cold and shiver after elective cesarean section.

Peri-operative hypothermia (body temperature below 36 ºC) is a cause of post-operative complications and patient discomfort. Immediately post-operatively such discomfort is due to increased pain and shivering. Patients say that their time in the recovery ward is very stressful and this is prolonged if they become cold (hypothermic)or shiver. Subsequently, patients can suffer with increased risk of infections and delayed discharge from hospital.

For patients (and their babies) having Cesarean sections it is important to start breast feeding as soon as possible, but being cold may delay this.

For some types of surgery measures are put in place to stop patients becoming cold and thereby reduce the number of problems. However this is not the case with patients undergoing Cesarean sections because the special blankets through which hot air is blown to keep them warm are inappropriate for mothers giving birth by Cesarean section as it would make it difficult for a mother to have good skin-to-skin contact with her new baby immediately after delivery - an important part in the bonding process.

A solution is to use a new warming mattress. This has been shown to be safe and effective with some types of surgery, but has not been tested in Cesarean sections.

In the investigators study,the investigators will warm a group of patients undergoing planned Cesarean section and compare them to an unwarmed group to see if there is any difference primarily in post-operative temperature. Secondarily, the investigators will also look for differences in total blood loss, incidence of blood transfusion, wound infection, shivering, the immediate health of the baby, time taken to become fit for discharge from recovery, length of hospital stay and time to breast-feeding.

DETAILED DESCRIPTION:
This project will be a randomised controlled trial comparing a warming mattress with current standard of care (no warming).

Prospective participants will be invited by letter and provided with a information booklet explaining the study and their rights. Informed consent will be taken in writing.

Patients will be randomised using a protocol created by the Trusts Clinical Investigations Research Unit who will use an Internet based randomisation system.

The researcher will not be blinded as it is not logistically feasible. The statistician analysing the results will be blinded to which group receives warming.

Study data will be collected manually on a standardised data collection sheet.

All enrolled patients will have their temperatures measured at specified times and will be observed for shivering. Data collection required to measure the primary outcomes will be complete by time of discharge from the recovery room. Data collection for secondary outcomes will be prospective and retrospective and will occur from time of anaesthesia through to one month after the procedure.

All patients will receive routine post-operative care.

To ensure any late complications are not missed we will interview the patients by phone one month after the date of their procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective (planned) caesarean section under spinal or combined spinal and epidural (CSE) anaesthesia will be eligible.

Exclusion Criteria:

* Exclusion criteria will be those who refuse, who are unable to fully understand the trial or are under 16 years of age when presenting for their Caesarean section.
* Those that are unable to understand for language issues are excluded with regret due to the difficulties of obtaining interpreters at the time of caesarean section, in recovery and once at home for the telephone interview. Waiting for additional interpretation may delay the clinical management of the patient and also the patient may not be able to convey questions or concerns about the study through mail, email or telephone prior to attending.
* Patients under 16 years of age will be excluded from the trial for reasons of consent. Although a patient less than 16 years of age may have Gillick competence and therefore have the capacity to consent to take part in this trial, as a minor their parents may have concerns leading them to refuse trial entry. Child birth in minors can be very stressful for the patient, family and clinical team and we are keen not to add to this for the purposes of a study.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Harper, MBBS, FRCA, Study Chair — BSUH NHS Trust, UK; Abhijoy Chakladar, MRCP, FRCA, Principal Investigator — BSUH NHS Trust, UK
Locations (1):
- Brighton and Sussex University Hospitals NHS Trust, Brighton, East Sussex, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February 2010- September 2012 Recruitment at preop assessment; consent on admission. Study location: obstetric ward and operating theatres
Pre-assignment Details: Entry into study phase on arrival in operating theatre. Final temperature readings to in the PACU
Groups:
- A Control: Standard Care: Control arm. Full standard care. No mattress warming. May receive warmed fluids if standard practise for clinician
- B Intervention: Warming Mattress: Warming mattress activated otherwise same management as Arm A.
  Warming with warming mattress: Reusable pressure relieving warming mattress. Principle use is to warm patients to prevent hypothermia peri-operatively.
  Inditherm Alpha systems, OTM1: 1900mm x 585mm
Period: Overall Study
Arm/Group | A Control: Standard Care | B Intervention: Warming Mattress
Started | 58 | 58
Completed | 58 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A Control: Standard Care | B Intervention: Warming Mattress | Total
Number analyzed (Participants) | 58 | 58 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (5.8) | 34.3 (5.9) | 34.0 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 58 | 116
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 58 | 58 | 116
Incidence IPH [Number; unit: participants] | 58 | 58 | 116

OUTCOME MEASURES:

1. Primary Outcome: This Study Intends to Investigate Whether an Electric Warming Mattress Can Reduce Post-operative Hypothermia (Defined as Body Temperature of Less Than 36.0ºC) in Patients Undergoing Planned Caesarean Section.
Description: IPH (body temperature of less than 36.0ºC)
Time Frame: On admission to recovery room - time variable, same day as procedure
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- A: Control Arm: Standard Care: Control arm. Full standard care. No mattress warming. May receive warmed fluids if standard practise for clinician
- B: Intervention: Warming Mattress: Warming mattress activated otherwise same management as Arm A.
  Warming with warming mattress: Reusable pressure relieving warming mattress. Principle use is to warm patients to prevent hypothermia peri-operatively.
  Inditherm Alpha systems, OTM1: 1900mm x 585mm
Arm/Group | A: Control Arm: Standard Care | B: Intervention: Warming Mattress
Number analyzed (Participants) | 58 | 58
participants | 58 [57 to 59] | 58 [57 to 59]

2. Primary Outcome: This Study Intends to Investigate Whether an Electric Warming Mattress Can Reduce the Incidence of Shivering in Patients Undergoing Planned Caesarean Section.
Description: Whether an electric warming mattress can reduce the incidence of shivering in patients undergoing planned Caesarean section. Shivering will be described according to severity on a scale of 1-4 where 1 is no shivering and 4 is uncontrolled shivering
Time Frame: From start of anaesthesia till discharge from the recovery room - time variable, same day as procedure
Reporting Status: Not Posted, anticipated posting 2020-07

3. Secondary Outcome: Differences in Total Blood Loss
Time Frame: At the end of the Caesarean section - time variable
Reporting Status: Not Posted

4. Secondary Outcome: Differences in Incidence of Blood Transfusion
Time Frame: From start of Caesarean section to discharge from hospital - times variable
Reporting Status: Not Posted

5. Secondary Outcome: Differences in Wound Infection Rates
Time Frame: From immediately post-operative till 1 month post procedure
Reporting Status: Not Posted

6. Secondary Outcome: Differences in Shivering (Severity and the Need for Treatment)
Time Frame: On admission to recovery room - time variable, same day as procedure
Reporting Status: Not Posted

7. Secondary Outcome: Differences in Immediate Health of Baby
Time Frame: At time of baby's birth - same day as Caesarean section
Reporting Status: Not Posted

8. Secondary Outcome: Differences in Time Taken for Mother to Become Fit for Discharge From Recovery
Time Frame: Time mother is ready for discharge from recovery room On admission to recovery room - time variable, same day as procedure
Reporting Status: Not Posted

9. Secondary Outcome: Differences in Length of Hospital Stay
Time Frame: Worked out reterospectively post-discharge from hospital patient notes
Reporting Status: Not Posted

10. Secondary Outcome: Differences in Time to Breast-feeding (if Mother Chooses to Breast Feed)
Time Frame: From time of admission to recovery room till breast feeding established On admission to recovery room - time variable, hopefully within 24hrs
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | A Control: Standard Care | B Intervention: Warming Mattress
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes